CLINICAL TRIAL: NCT07284992
Title: Total Neoadjuvant Treatment With Short-course Radiotherapy Versus Long-course Radiotherapy Followed by PD-L1 Inhibitor Plus Capecitabine-Oxaliplatin in Patients With Locally Advanced Rectal Cancer: a Multi-centres, Open-label, Phase 2, Randomized Controlled Trial
Brief Title: SCRT VS LCRT Followed by PD-L1 Inhibitor Plus CAPEOX as TNT in Patients With LARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Feng Tian, Associate Professor, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPRING03
Record Dates: First submitted 2025-11-18; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Rectal Cancer; Advanced Stage Colorectal Cancer; Radiotherapy
Keywords: Immune checkpoint inhibitors; Adebrelimab Injection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Radiotherapy protocol: 5 × 5Gy short-term radiotherapy (D1-5 in the first week) Immunotherapy regimen: Adebrelimab 1200 mg or 20 mg/kg, IV., administered on the first day of each chemotherapy cycle.
  Chemotherapy regimen: capox regimen:
  Oxaliplatin 130 mg/m2 IV D1 Capecitabine 1000 mg/m2 Po bid D1 ～ 14 Repeat every 3 weeks for 6 cycles The curative effect was evaluated 2-3 weeks after the completion of 6 cycles of chemotherapy. According to whether the CCR (clinical complete remission) was achieved, TME surgery was required if the CCR was not achieved; If CCR is achieved, TME operation can be performed according to the wishes of the patients. Local resection or observation through anal surgery requires close follow-up to explore the effectiveness and safety of the scheme.
  Interventions: Combination Product: short-term radiotherapy combined with Adebrelimab and capox
- Group 2 (Experimental): Radiotherapy regimen: long-term radiotherapy 1.8 × 25-28Gy, oral capecitabine in the same period: the standard dose is 825mg/m2, twice a day [total dose 1650mg/(M2 · d)], oral radiotherapy day, 5 days a week.
  Immunotherapy regimen: Adebrelimab 1200 mg or 20 mg/kg, IV., administered on the first day of each chemotherapy cycle.
  Chemotherapy regimen: capox regimen:
  Oxaliplatin 130 mg/m2 IV D1 Capecitabine 1000 mg/m2 Po bid D1 ～ 14 Repeat every 3 weeks for 6 cycles The curative effect was evaluated 2-3 weeks after the completion of 6 cycles of chemotherapy. According to whether the CCR (clinical complete remission) was achieved, TME surgery was required if the CCR was not achieved; If CCR is achieved, TME operation can be performed according to the wishes of the patients. Local resection or observation through anal surgery requires close follow-up to explore the effectiveness and safety of the scheme.
  Interventions: Combination Product: long-term radiotherapy combined with Adebrelimab and capox

INTERVENTIONS:
Combination Product: short-term radiotherapy combined with Adebrelimab and capox — Radiotherapy protocol: 5 × 5Gy short-term radiotherapy (D1-5 in the first week) Immunotherapy regimen: Adebrelimab 1200 mg or 20 mg/kg, IV., administered on the first day of each chemotherapy cycle.
  Chemotherapy regimen: capox regimen:
  Oxaliplatin 130 mg/m2 IV D1 Capecitabine 1000 mg/m2 Po bid D1 ～ 14 Repeat every 3 weeks for 6 cycles The curative effect was evaluated 2-3 weeks after the completion of 6 cycles of chemotherapy. According to whether the CCR (clinical complete remission) was achieved, TME surgery was required if the CCR was not achieved; If CCR is achieved, TME operation can be performed according to the wishes of the patients. Local resection or observation through anal surgery requires close follow-up to explore the effectiveness and safety of the scheme.
  Other Names: Adebrelimab; CAPOX
  Arms: Group 1
Combination Product: long-term radiotherapy combined with Adebrelimab and capox — Radiotherapy regimen: long-term radiotherapy 1.8 × 25-28Gy, oral capecitabine in the same period: the standard dose is 825mg/m2, twice a day [total dose 1650mg/(M2 · d)], oral radiotherapy day, 5 days a week.
  Immunotherapy regimen: Adebrelimab 1200 mg or 20 mg/kg, IV., administered on the first day of each chemotherapy cycle.
  Chemotherapy regimen: capox regimen:
  Oxaliplatin 130 mg/m2 IV D1 Capecitabine 1000 mg/m2 Po bid D1 ～ 14 Repeat every 3 weeks for 6 cycles The curative effect was evaluated 2-3 weeks after the completion of 6 cycles of chemotherapy. According to whether the CCR (clinical complete remission) was achieved, TME surgery was required if the CCR was not achieved; If CCR is achieved, TME operation can be performed according to the wishes of the patients. Local resection or observation through anal surgery requires close follow-up to explore the effectiveness and safety of the scheme.
  Other Names: Adebrelimab; CAPOX
  Arms: Group 2

SUMMARY:
This is a multicenter, cohort, prospective study to evaluate the efficacy and safety of Adebrelimab combined with radiotherapy and chemotherapy as preoperative neoadjuvant therapy for patients with locally advanced rectal cancer. In the study, all subjects who meet the inclusion criteria will enter the short-term radiotherapy queue and the long-term radiotherapy queue at the ratio of 1:1. The short-term radiotherapy queue plans to receive Adebrelimab combined with short-term radiotherapy (5*5Gy) and Capox chemotherapy as neoadjuvant therapy. The long-term radiotherapy queue plans to receive Adebrelimab combined with long-term radiotherapy (1.8gy × 25-28 times) and capox chemotherapy as neoadjuvant therapy. The TME surgery will be performed 2-3 weeks after the last neoadjuvant therapy is completed. If the surgery cannot be performed within the time window specified in the plan (such as delayed adverse reactions, etc.), the researcher will conduct the surgery according to the patients' requirements.The actual clinical conditions of the subjects were comprehensively considered.

ELIGIBILITY:
Inclusion Criteria:

* 1. sign written informed consent before implementing any test related process;
* 2. Patients diagnosed as rectal adenocarcinoma by primary biopsy and histopathological examination;
* 3. patients with CT stage ≥ T3 or CN stage N1+, M0 or EMVI (+) or MRF (+) or suspected lateral lymph node metastasis (>5mm) who are judged by imaging and colonoscopy to be operable and need neoadjuvant therapy.
* 4. according to imaging and colonoscopy, the main body of the tumor was located ≤ 10cm from the anal edge;
* 5. patients with tumor mismatch repair/microsatellite instability (MMR/MSI) status as MSS;
* 6. according to the criteria for evaluating the efficacy of solid tumors (RECIST version 1.1), at least one lesion can be measured by imaging;
* 7. the patient has not received any anti-tumor treatment in the past, including but not limited to surgery, radiotherapy, chemotherapy, immunotherapy, targeted therapy, etc;
* 8. ECoG score: 0-1;
* 9. sufficient organ function, the subject shall meet the following laboratory indicators:

  1. The absolute value of neutrophils (ANC) ≥ 1.5x109/l without granulocyte colony stimulating factor in the past 14 days.
  2. Platelets ≥ 100 × 109/l without blood transfusion in recent 14 days.
  3. Hemoglobin>9g/dl without blood transfusion or use of erythropoietin in recent 14 days;
  4. Total bilirubin ≤ 1.5 × upper limit of normal value (ULN);
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) in ≤ 2.5 × ULN
  6. Serum creatinine ≤ 1.5 × ULN and creatinine clearance rate (calculated by Cockcroft Gault formula) ≥ 60 ml/min;
  7. Good coagulation function was defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN;
  8. Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is beyond the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
  9. Myocardial enzyme spectrum is within the normal range (for example, simple laboratory abnormalities that are not clinically significant according to the comprehensive judgment of the researcher are also allowed to be included in the group)
* 10. female subjects of childbearing age should receive urine or serum pregnancy test within 3 days before receiving the first study drug administration (the first day of the first cycle) and the result is negative. If the result of urine pregnancy test cannot be confirmed as negative, blood pregnancy test is required. Women of non reproductive age were defined as having been postmenopausal for at least 1 year, or having undergone surgical sterilization or hysterectomy; If there is a risk of pregnancy, all subjects (male or female) need to take contraceptive measures with an annual failure rate of less than 1% during the whole treatment period until 120 days after the last study drug administration (or 180 days after the last chemotherapy drug administration).

Exclusion Criteria:

* 1. patients diagnosed with other malignant tumors and not cured within 5 years before the first administration (excluding skin basal cell carcinoma, skin squamous cell carcinoma, and/or cancer in situ after radical resection);
* 2. Patients with advanced rectal cancer with distant metastasis;
* 3. currently participating in intervention clinical research treatment, or having received other research drugs or used research instruments within 4 weeks before the first administration;
* 4. have previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that stimulate or synergistically inhibit T cell receptors (e.g., CTLA-4, OX-40, CD137);
* 5. have received systemic treatment with Chinese patent medicine with anti-tumor indications or drugs with immunomodulatory effect within 2 weeks before the first administration;
* 6. active autoimmune diseases requiring systemic treatment (such as the use of disease relieving drugs, glucocorticoids or immunosuppressants) occurred within 2 years before the first administration. Replacement therapy (such as thyroxine, insulin or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) is not considered as systemic therapy;
* 7. the patients were receiving systemic glucocorticoid therapy (excluding local glucocorticoids via nasal spray, inhalation or other routes) or any other form of immunosuppressive therapy within 14 days before the first administration of the study; Note: it is allowed to use physiological doses of glucocorticoids (≤ 10 mg/day of prednisone or equivalent drugs); In the absence of active autoimmune diseases, inhaled or topical steroid and prednisone dose>10mg/day or equivalent dose of adrenocortical hormone are allowed to replace;
* 8. known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* 9. those who are known to be allergic to the study drug adebaylimab and the active ingredients or excipients of combined chemotherapy drugs;
* 10. have not fully recovered from the toxicity and/or complications caused by any intervention measures before starting treatment (i.e. ≤ grade 1 or reaching the baseline, excluding fatigue or hair loss);
* 11. known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
* 12. untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected is greater than the upper limit of normal value in the laboratory of the research center);

Note: hepatitis B subjects who meet the following criteria can also be enrolled:

1. HBV viral load<1000 copies/ml (200 iu/ml) before the first administration. Subjects should receive anti HBV treatment during the whole study chemotherapy drug treatment to avoid virus reactivation
2. For subjects with anti HBC (+), HBsAg (-), anti HBS (-) and HBV viral load (-), preventive anti HBV treatment is not required, but virus reactivation needs to be closely monitored

   * 13. active HCV infected subjects (HCV antibody positive and HCV-RNA level higher than the detection limit);
   * 14. inoculate live vaccine within 30 days before the first administration (cycle 1, day 1); Note: it is allowed to receive inactivated virus vaccine for injection against seasonal influenza within 30 days before the first administration; However, live attenuated influenza vaccines administered intranasal are not allowed.
   * 15. pregnant or lactating women;
   * 16. there are any serious or uncontrollable systemic diseases, such as:

1) The resting ECG has significant abnormalities in rhythm, conduction or morphology, and the symptoms are serious and difficult to control, such as complete left bundle branch block, heart block above grade II, ventricular arrhythmia or atrial fibrillation; 2) Unstable angina pectoris, congestive heart failure, chronic heart failure with NYHA classification ≥ 2; 3) Myocardial infarction occurred within 6 months before enrollment; 4) Blood pressure control was not ideal (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg); 5) There was a history of non infectious pneumonia requiring glucocorticoid treatment within 1 year before the first administration, or there was currently clinically active interstitial lung disease; 6) Active pulmonary tuberculosis; 7) Active or uncontrolled infection requiring systemic treatment; 8) There were clinically active diverticulitis, abdominal abscess and gastrointestinal obstruction; 9) Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis; 10) Poor control of diabetes mellitus (FBG>10mmol/L); 11) The urine routine showed that the urine protein was ≥++, and it was confirmed that the 24-hour urine protein quantitation was more than 1.0 G; 12) Patients with mental disorders and unable to cooperate with treatment;

* 17. for those who have a history of uncontrolled epilepsy, central nervous system disease or mental disorder, the clinical severity may hinder the signing of informed consent or affect the patient's compliance with oral drugs according to the judgment of the investigator; The medical history or disease evidence, abnormal treatment or laboratory test values that may interfere with the test results, prevent the subjects from participating in the whole process of the study, or the researchers believe that there are other potential risks that are not suitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
CR rate | From enrollment to the end of surgery,assessed up to 6 months
  pathological complete remission rate (PCR) and clinical complete remission rate (CCR)

SECONDARY OUTCOMES:
partial remission rate (PR) | The evaluation time from enrollment to the first efficacy evaluation is up to 3 months
  the total diameter of all measurable target lesions is ≥ 30% lower than the baseline
Objective response rate (ORR) | The evaluation time from enrollment to the first efficacy evaluation is up to 3 months
  Proportion of subjects defined as complete remission (CR) and partial remission (PR) in total subjects
Major Pathological Response Rate (MPR) | From enrollment to the end of surgery,assessed up to 6 months
  Major Pathological Response Rate (MPR)
R0 resection rate | From enrollment to the end of surgery,assessed up to 6 months
  There is no visible tumor residue in the body, and no residual tumor cells are found under the pathological microscope
2-year DFS rate | The longest follow-up time was 2 years from enrollment to disease progression
  2-year progression free survival rate
3-year OS rate | The longest follow-up time was 3 years from enrollment to death from any cause
  3-year OS rate

CONTACTS AND LOCATIONS:
Overall Officials: Changqing Jing, Professor, Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided